CLINICAL TRIAL: NCT02877966
Title: Evaluation of the Effects of a Stoichiometric Mixture of Amino Acids (Amixea) on Lean Body Mass and Muscle Strengh of Patients With Unresectable Advanced Non-small Cell Lung Cancer: a Randomized, Double Blind, Placebo-controlled, Multicenter Study
Brief Title: Evaluation of the Effects of a Mixture of Amino Acids (Amixea) on Lean Body Mass and Muscle Strengh of Patients With Unresectable Advanced Non-small Cell Lung Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of Trial Sponsor
Sponsor: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HF03-14-37
Record Dates: First submitted 2016-01-27; First posted 2016-08-25 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Cancer Patients With Cachexia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Amixea- patented stoechiometrical mixture of EAA & AA
  Interventions: Dietary Supplement: Amixea
- Arm B (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Amixea — Amixea is a mixture of amino acids. It consists mainly of essential amino acids (EAA) that cannot be synthesized de novo by the organism, and therefore must be supplied in its diet.
  Arms: Arm A
Other: Placebo
  Arms: Arm B

SUMMARY:
The primary objectives of this study are to evaluate the effects of an amino acid mixture (Amixea) on the body composition as assessed by DXA, and on QMVC as assessed by strain gauge, in advanced NSCLC patients, compared to placebo, after 10 weeks of treatment.

Secondary objectives are to evaluate the activity of Amixea on the degree of protein synthesis, on the nutritional risk and status and quality of life in advanced NSCLC patients, compared to placebo, after 10 weeks of treatment. In a small subsample, body composition will be evaluated opportunistically from clinically available CT scans.

Adherence to, and patient satisfaction of treatment will be evaluated as exploratory objectives of this study. Finally, the overall safety and product tolerability will be evaluated.

DETAILED DESCRIPTION:
Most cancer patients experience weight loss at some time as their disease progresses. The resulting malnutrition increases risk of treatment complication and may lead to poor treatment response and/or tolerance, reduced quality of life and poor survival. The prevalence of malnutrition in cancer patients is thought to be as high as 80%, but reports vary with cancer location and stage, treatment history, clinical setting and assessment criteria.

Weight loss with cachexia is a common presenting sign in NSCLC, representing a great concern for many patients and their families. At this regard, NSCLC cachexia is worth of particular investigation because of the prevalence of the disease, the frequency with which it is associated with weight loss and the prognostic implications of weight loss for these patients.

Weight stabilization may be the most optimistic outcome to be expected in patients with cachexia and is still beneficial, as weight-losing patients with cancer cachexia who stabilize their weight have a greater quality of life and survival then those who continue to lose weight.

It is, in fact, well-known that cachexia increases cancer-related mortality and has devastating effects on quality of life.Randomized controlled trial data indicate that early palliative care improves quality of life and depressive symptoms and may extend survival in advanced NSCLC compared with standard care.

In particular, it has been observed that conventional nutritional supplements are not or only partly successful in inducing protein accretion in advanced cancer, suggesting an attenuated anabolic response. To prevent muscle wasting and its deleterious consequences, generating an anabolic response is crucial. Dietary essential amino acids (EAA) have anabolic properties in other wasting diseases, however data in advanced cancer are lacking.

Previous studies have analyzed patients with chronic obstructive pulmonary disease with cachexia or skeletal muscle dysfunction and have demonstrated quadriceps weakness in one-third of COPD patients attending hospital respiratory outpatient services.

An accurate and rapid evaluation of muscle strength which may identify patients with muscle weakness could be of crucial importance in a prompt and specific intervention in prescribing an adequate support therapy.

Starting from these assumptions, the main objectives of this study are to evaluate the effects of an amino acids mixture (Amixea) on the body composition by dual-energy x-ray absorptiometry (DXA), a bone mineral densitometer, and on quadriceps maximal voluntary contraction force (QMVC) in advanced NSCLC patients, compared to placebo, after 10 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Females and males at least 18 years of age.
2. Stage III or IV unresectable NSCLC (documented histologic or cytologic diagnosis according to AJCC Cancer Staging).
3. On or planned first line chemotherapy or targeted therapies.
4. ECOG performance status ≤ 2.
5. Estimated life expectancy of > 6 months at the time of screening.
6. Adequate hepatic function, defined as aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤5 x upper limit of normal (ULN).
7. Adequate renal function, defined as creatinine ≤2 x ULN, or calculated creatinine clearance >30 ml/minute.
8. Must be willing and able to give signed informed consent and, in the opinion of the Investigator, to comply with the protocol tests and procedures.

   -

Exclusion Criteria:

1. Other forms of lung cancer (eg, small cell, mesothelioma)
2. Women who are pregnant or breast-feeding
3. Known HIV, hepatitis (B & C), or active tuberculosis
4. Had major surgery (central venous access placement and tumor biopsies are not considered major surgery) within 4 weeks prior to randomization. Patients must be well recovered from acute effects of surgery prior to screening. Patients should not have plans to undergo major surgical procedures during the treatment period.
5. Patients undergoing curative radiation therapy.
6. Patients on treatment with levodopa.
7. Patients unable to readily swallow. Patients with severe gastrointestinal disease (including esophagitis, gastritis, malabsorption, or obstructive symptoms) or intractable or frequent vomiting are excluded.
8. Patients with active, uncontrolled infection.
9. Patients with uncontrolled diabetes mellitus.
10. Patients with untreated, clinically relevant hypothyroidism.
11. Patients with known or symptomatic brain metastases.
12. Patients receiving parenteral nutrition (either total or partial).
13. Other clinical diagnosis, ongoing or intercurrent illness that in the Investigator's opinion would prevent the patient's participation.
14. Use of other investigational drug(s) within 30 days before study entry or during the study.

    -

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
effects of an amino acid mixture (Amixea) on the body composition | 10 weeks of treatment
  Lean Body Mass determination with DXA scan and Maximal Voluntary Contraction Force using dynamometer (strain gauge)

SECONDARY OUTCOMES:
to evaluate the nutritional risk and status and quality of life in advanced NSCLC patients | 10 weeks of treatment
  Nutritional status and risk using the scored Patient-Generated Subjective Global Assessment (PG-SGA) tool
overall safety and product tolerability | 10 weeks of treatment
  Number and typology of adverse events (AEs), Physical examination and vital signs, Product tolerability

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Bond University-Department of Nutrition & Dietetics, Robina
  - Gold Coast University Hospital, Southport
  - Princess Alexandra Hospital, Woolloongabba

IPD SHARING:
Plan to Share IPD: No